CLINICAL TRIAL: NCT03930927
Title: Evaluation of the Re-mineralizing Effect of Biomimetic Self-Assembling Peptides in Post Orthodontic White Spot Lesions Compared to Fluoride-Based Delivery Systems
Brief Title: Effect of Self Assembling Peptide on White Spot Lesion
Acronym: regeneration
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Raneen Ahmed (Other)
Responsible Party: Sponsor-Investigator, Raneen Ahmed, assistant lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1998
Record Dates: First submitted 2019-04-19; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: White Spot Lesion of Tooth
MeSH Terms: interventions — P11-4 peptide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self Assembling peptide (Experimental): intervention
  Interventions: Drug: Self Assembling peptide; Drug: remineralizing agent
- Fluoride (Experimental): Comparator
  Interventions: Drug: Self Assembling peptide; Drug: remineralizing agent

INTERVENTIONS:
Drug: Self Assembling peptide — enamel regeneration
  Other Names: Curodont
Drug: remineralizing agent — enamel regeneration
  Other Names: floride

SUMMARY:
During re-mineralization of white spot lesion, Will biomimetic self-assembling peptides improve the re-mineralizating effect of the post orthodontic white spot lesion compared to fluoride-based delivery systems?

DETAILED DESCRIPTION:
Conservative dentistry no longer prefers the "drill and fill" concept and advocates reversal of lesions via remineralization. . Remineralization is the process of restoring minerals - again, in the form of mineral ions - to the hydroxyapatite latticework structure. It is three-dimensional, and the lost ions must be replaced with ions having the exact same shape, size and the same electrical charge as those lost from the lattice.

Fluoride and self-assembling peptides have been used as adjuncts to enhance remineralization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with post orthodontic white spot lesion.
* Patients with good oral hygiene.
* Patients with good general health.
* Cooperative patients.
* Subjects who signed the informed consent.

Exclusion Criteria:

* Patients with tetracycline pigmentation and dental fluorosis.
* Enamel cavitation.
* Disable patient.
* patient with any systemic disease or severe medical complications.

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Remineralizing process | 6 months
  using DIAGNOpen.

SECONDARY OUTCOMES:
Visual assessment | 6 months
  using ICDAS II

IPD SHARING:
Plan to Share IPD: Undecided